CLINICAL TRIAL: NCT00284037
Title: Improvement in Baroreflex Sensitivity in OSAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nagoya University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NU-06-A-0003
Record Dates: First submitted 2006-01-27; First posted 2006-01-31 (Estimated); Last update posted 2006-01-31 (Estimated); Status verified 2005-05

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: obstructive sleep apnea,; baroreceptors
MeSH Terms: conditions — Sleep Apnea, Obstructive

INTERVENTIONS:
Device: continuous positive airway pressure therapy

SUMMARY:
Individuals with obstructive sleep apnea syndrome (OSAS) are at high risk for cardiovascular morbidity and mortality. The effect of long-term nocturnal therapy with continuous positive airway pressure (CPAP) on daytime baroreflex sensitivity (BRS), a predictor of cardiac death, was investigated in OSAS patients.

ELIGIBILITY:
Inclusion Criteria:

* obstructive sleep apnea syndrome

Exclusion Criteria:

* diabetes mellitus, chronic obstructive lung disease, coronary or valvular heart disease, congestive heart failure, renal failure, or endocrine dysfunction. Moreover, none of them were taking b-blockers, vasodilators, or inotropic agents at the time of enrollment in the study.

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Mitsuhiro Yokota, MD.PhD, Study Chair — Department of Cardiovascular Genome Science, Nagoya University School of Medicine, Nagoya, Aichi, Japan
Locations (1):
- Nagoya University of Health Sciences, Nagoya, Japan